CLINICAL TRIAL: NCT04025398
Title: REHABILITUS: a New Cognitive Remediation Tool for Adults With Intellectual Deficiency With Behavioral Disorders
Brief Title: A Computer-based Cognitive Remediation Program for Adults With Intellectual Disability
Acronym: REHABILITUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-A00179-48
Record Dates: First submitted 2019-07-17; First posted 2019-07-18 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Intellectual Disability
MeSH Terms: conditions — Intellectual Disability | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: It's a study prospective, randomized, multicenter and controlled which compares two groups of people adults: group to remediation Réhabilitus versus group Control.
Who Masked: Outcomes Assessor
Masking Description: Blindness of the psychologist for the secondary judgment criteria.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- REHABILITUS (Experimental): Réhabilitus is a cognitive remediation program focused on the functions of attention and visuospatial that is to say that can move in space, to perceive objects of our environment and organize them, to mentally imagine a physically absent operation object very involved in social behavior, in order to limit the presence of behavioral disorders among adults with intellectual disabilities.
  Interventions: Behavioral: Cognitive remediation program
- CONTROL GROUP (Active Comparator): The control group involves manual activities and research computer information.
  Interventions: Behavioral: Control group

INTERVENTIONS:
Behavioral: Cognitive remediation program — Comparison between a cognitive remediation program (REHABILITUS) (group 1) and a training group of manual activities (group 2)
  Arms: REHABILITUS
Behavioral: Control group — Comparison between a cognitive remediation program ("Réhabilitus") (group 1) and a training group of manual activities (group 2)
  Arms: CONTROL GROUP

SUMMARY:
Adults with intellectual disabilities have great difficulty in adapting to social situations and relationships. Cognitive impairment associated with intellectual disability are important factors to understand their difficulties in processing social information. In the field of recognition of facial emotions in particular, basic cognitive processes such as visuospatial and attentional functions, are heavily involved. Cognitive remediation is a management tool widely used by practitioners to help patients who experience cognitive difficulties. Currently, no program can meet specific and validated the problems are adults with intellectual disabilities manner in their daily functioning

DETAILED DESCRIPTION:
Réhabilitus is a remediation program focused on attentional functions and visuospatial, to limit the presence of behavioral disorders among adults with intellectual disabilities. The main objective is to validate the effectiveness of Réhabilitus program on behavioral disorders in adults with intellectual disabilities without autism spectrum disorder associated.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 45 inclusive;
* Behavioral disorders corresponding to a total score on the ABC scale > 15
* Presence of a family caregiver (parent, friend) or professional (reeducator, professional of the medico-social sector) stakeholder of the project;
* Diagnosis of mild to moderate intellectual disability (assessed by WAIS-IV battery and VABS-II less than 3 years ago;
* French or secondary mother tongue;
* Psychoactive treatment unchanged during the month prior to inclusion;
* Adult or legal representative who has given written and informed consent to participate in the study. By default, the adult's oral agreement will be collected (as well as the written consent of the legal representative);
* Affiliation to the social security scheme or beneficiary of such a scheme.

Exclusion Criteria:

* Neurological disorders of vascular, infectious or neurodegenerative origin;
* Taking medications for general medical purposes with a neurological or psychiatric impact (eg corticosteroids);
* Simultaneous participation in any other cognitive remediation program targeting attentional, visuospatial and social cognition;
* Refusal of participation of the person and/or his/her legal representative;
* Not family or professional caregiver;
* Presence of Autistic Spectrum Disorders (evaluated by ADOS and ADI if necessary according to the assessment of the investigator)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 116 (Estimated)
Dates: Start 2020-06-17 (Actual); Primary Completion 2026-06-17 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in sub-score hyperactivity / non compliance on Aberrant Behavior Checklist scale | 6 months
  Aberrant Behavior Checklist scale (ABC) The ABC scale [20] is a 58-item scale for people close to the autistic person. Scores are distributed in five subscale: irritability, agitation, crying; of lethargy and social withdrawal; stereotyped behaviors; hyperactivity; inappropriate language.

SECONDARY OUTCOMES:
This measure is repeated at the end of the intervention to highlight the impact of the " Cognitus and Me " program, and 6 months later to investigate the possible long-lasting effects of the benefits | 6 months
  ABC scale (Irritability and social withdrawal)
Change from baseline in facial emotion recognition task | 6 months
  Facial Emotions Recognition Task (TREF)
Change from baseline in attentional functions | 6 months
  Sustained Attention on LEITER-3 Battery Attention scales and memory - forward memory, reverse memory, sustained attention, divided attention, non-verbal stroop.

CONTACTS AND LOCATIONS:
Overall Officials: DEMILY CAROLINE, MD Ph, Principal Investigator — Centre Hospitalier le Vinatier
Locations (1):
- Hopital Vinatier, Lyon, Auvergne-Rhône-Alpes, France

IPD SHARING:
Plan to Share IPD: No